CLINICAL TRIAL: NCT04910360
Title: Examining the Genetic Predisposition of Individuals Who Aggravated by Embolism in COVID-19 Positive Patients
Brief Title: Embolism in COVID-19 Positive Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Semiha Orhan, Medical doctor, Afyonkarahisar Health Sciences University
Other Study IDs: 2021-1
Record Dates: First submitted 2021-05-31; First posted 2021-06-02 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: COVID-19 Pneumonia; Embolism; Genetic Predisposition
Keywords: thrombophilia; genetic factors; COVID-19
MeSH Terms: conditions — Embolism; Genetic Predisposition to Disease; Thrombophilia; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 3 ml blood samples and extracted DNA from blood samples are stored.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICU patients with severe COVID-19 pneumonia: Without using any intervention, this group has been included in the study to research certain genetic dispositions determining the severity of the COVID-19 pneumonia
- Random population: This group has been included as a control group to compare the genetic predisposition of ICU patients with severe COVID-19 pneumonia with the normal population.

SUMMARY:
Covid-19 outbreak has caused death of millions of people because of not only the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection itself but also infection dependent complications. Abnormalities in thrombotic events leads to some of these complications which eventually result in emboli. The endothelial damage caused by the virus interacting with ACE2 on the host cells leads to the activation of coagulation cascade. Accumulation of byproducts of the cascade might have some roles in embolism inducing risk of organ damage, other life-threatening problems, and even death. To enlighten the factors triggering embolism, the investigators have focused on genetic changes such as polymorphisms and mutations in certain genes in DNA samples coming from intensive care unit (ICU) patients.

DETAILED DESCRIPTION:
This study has conducted to find the possible links between genetic make up of ICU patients with severe Covid-19 and embolism. 13 polymorphisms and mutations that the investigators targeted are located on Factor II, Factor V, Factor XIII, MTHFR, angiotensin converting enzyme (ACE), endothelial cell protein C receptor (EPCR), and FGB. The investigators have found significant changes in the mutant allele frequencies in most of the factors.

The main workflow to study a point change on DNA sequence begins with DNA isolation from a biological material. In this case, we received blood samples in ethylenediaminetetraacetic acid (EDTA) tubes from ICU patients with severe Covid-19. The investigators hypothesis claims that genetic factors triggering thrombotic events might increase the severity of the diseases by inducing the risk of emboli.

After DNA isolation, desired loci on DNA were amplified via Polymerase Chain Reaction (PCR). Amplicons including the mutations and polymorphisms need to be purified before next generation sequencing (NGS).

The investigators analyze the data using Integrative Genomics Viewer (IGV) program and check the genetic profile (wt, het, mut). Some of the changes are meaningful by themselves while some other need to be considered as combinations. Compound heterozygosity and diagnosis for thrombophilia require cooccurrence of the changes.

To compare allelic frequencies, the investigators include the average of the data coming from more than 2000 individuals with no know thrombophilia cases. In the investigators focus cohort, the investigators have the data of 47 Covid-19 patients in ICU.

ELIGIBILITY:
Inclusion Criteria:

* being tested positive for Covid-19
* ICU patients developing severe pneumonia upon Covid-19 infection

Exclusion Criteria:

* previously tested positive for genetic factors increasing thrombosis risk
* ICU patients developing severe emboli regardless of Covid-19 infection

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Groups were assigned to determine the genetic factors that explain severity of COVID-19 infections. These genetic factors play role in thrombotic events in the body.
  Case group involves ICU patients with emboli that suffer from severe COVID-19. The investigators expect to see some deviations from normal population regarding the mutations and polymorphisms related to thrombophilia. Control group is normal population representing the normal allelic frequencies of the determinant genetic factors.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-05-08 (Actual); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Changes in allelic frequencies in predetermined loci which are known to be related with thrombosis | 15.03.2021- 30.04.2021
  In the first 28 samples the investigators received, we expected a predictive result revealing the genetic background and embolism in Covid-19. Deviations from allelic frequencies of healthy population regarding some of the factors will support the hypothesis of the study.
An increase in thrombophilia cases in the study group | 01.05.2021- 20.05.2021
  Thrombophilia is a complex state with the contribution of several factors. Clinical picture and the mutations enable the diagnosis. With an expanded study group consisting of 47 patients, we determined the patients with thrombophilia.

CONTACTS AND LOCATIONS:
Overall Officials: Serdar Ceylaner, Assoc. Prof., Study Director — INTERGEN Genetics and Rare Diseases Diagnosis Research & Application Center
Locations (1):
- INTERGEN Genetics and Rare Diseases Diagnosis Research & Application Center, Ankara, Cankaya, Turkey (Türkiye)